CLINICAL TRIAL: NCT02781792
Title: A Randomized Feasibility Study Evaluating Temozolomide Chronotherapy for High Grade Glioma
Brief Title: Temozolomide Chronotherapy for High Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201605081
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Glioma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Temozolomide morning (Experimental): * Temozolomide will be given as per standard of care. Typical dosing is 150 to 200 mg/m^2 on Days 1 through 5 of a 28-day treatment cycle. Patients will be randomized to take their temozolomide doses in the morning (before 10:00).
  * FACT-Br quality of life at baseline, at the beginning of each cycle of chemotherapy, and 1 month after the final chemotherapy treatment
  Interventions: Drug: Temozolomide; Other: Functional Assessment of Cancer Therapy - Brain; Other: ActTrust Condor Instrument Watch
- Arm 2: Temozolomide evening (Experimental): * Temozolomide will be given as per standard of care. Typical dosing is 150 to 200 mg/m2 on Days 1 through 5 of a 28-day treatment cycle. Patients will be randomized to take their temozolomide doses in the evening (after 20:00).
  * FACT-Br quality of life at baseline, at the beginning of each cycle of chemotherapy, and 1 month after the final chemotherapy treatment
  Interventions: Drug: Temozolomide; Other: Functional Assessment of Cancer Therapy - Brain; Other: ActTrust Condor Instrument Watch

INTERVENTIONS:
Drug: Temozolomide — -Given standard of care
  Other Names: Temodar
Other: Functional Assessment of Cancer Therapy - Brain — * 23-item questionnaire that can be completed in 5 to 10 minutes with little or no assistance in patients who are not neurologically incapacitated. This brain subscale is usually used along with the core (general) questionnaire [2] that includes 27 items.
  * Patients rate all 5 items using a five-point Likert scale ranging from 0 "not at all" to 4 "very much." Overall, higher ratings suggest higher QOL. Items are totaled to produce the following subscales, along with an overall QOL score: physical well-being (7 items); social/family well-being (7 items); emotional well-being (6 items); functional well-being (7 items); and concerns relevant to patients with brain tumors (23 items)
  * The sleep portion of this questionnaire consists of 17 questions about sleeping patterns and the ability to rate severity of insomnia.
  Other Names: FACT-Br
Other: ActTrust Condor Instrument Watch — -Will be required to wear 24 hours per day and will only be removed at specified data collection time points

SUMMARY:
Temozolomide (TMZ) is the chemotherapy drug approved by the FDA to increase survival in glioblastoma (GBM) patients beyond surgical resection and radiation therapy alone. Give its activity in astrocytomas, TMZ is commonly used in grade III anaplastic astrocytoma (AA) as well. Both grade III AA and grade IV GBM are high grade gliomas (HGG). The short half-life of this drug and known oscillations in DNA damage repair make it an ideal candidate for chronotherapy.

Chronotherapy is the improvement of treatment outcomes by minimizing treatment toxicity and maximizing efficacy through delivery of a medication according to the timing of biological rhythms within a patient. Chronotherapy has improved outcomes through the reduction of side effects and increase in anti-tumor activity for a variety of cancers, but has never been applied to the treatment of gliomas.

Based on the preliminary preclinical data for chronotherapeutic TMZ treatment of intracranial glioma xenografts and the success of chronotherapy in the treatment of other cancers, the investigators hypothesize that the timing of TMZ treatment will alter its efficacy and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and recurrent high grade gliomas (WHO grades III & IV) and high risk WHO grade II gliomas who are to begin treatment with monthly high dose temozolomide therapy.
* Scheduled to receive adjuvant temozolomide therapy after having completed concurrent temozolomide and radiation therapy.
* At least 18 years of age.
* Karnofsky performance status ≥ 60%
* Ability to understand and willingness to sign an IRB approved written informed consent document

Exclusion Criteria:.

-Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milan Chheda, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Damato AR, Katumba RGN, Luo J, Atluri H, Talcott GR, Govindan A, Slat EA, Weilbaecher KN, Tao Y, Huang J, Butt OH, Ansstas G, Johanns TM, Chheda MG, Herzog ED, Rubin JB, Campian JL. A randomized feasibility study evaluating temozolomide circadian medicine in patients with glioma. Neurooncol Pract. 2022 Jan 31;9(3):193-200. doi: 10.1093/nop/npac003. eCollection 2022 May. PMID 35601970
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Temozolomide Morning: -Temozolomide will be given as per standard of care. Typical dosing is 150 to 200 mg/m^2 on Days 1 through 5 of a 28-day treatment cycle. Patients will be randomized to take their temozolomide doses in the morning (before 10:00).
- Arm 2: Temozolomide Evening: -Temozolomide will be given as per standard of care. Typical dosing is 150 to 200 mg/m2 on Days 1 through 5 of a 28-day treatment cycle. Patients will be randomized to take their temozolomide doses in the evening (after 20:00).
Period: Overall Study
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
Started | 22 | 20
Completed | 17 | 15
Not Completed | 5 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Hospice | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.59 (12.35) | 53.05 (17.52) | 55.95 (15.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 10 | 14 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 21 | 18 | 39
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 0 | 2
  White | 19 | 18 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Patient Treatment Compliance as Measured by Number of Participants Who Were at Least 80% Compliance With Assigned Administration Time
Description: Compliance is defined as no more than one of five doses of temozolomide per cycle taken outside of the assigned administration time.
Time Frame: Through completion of treatment (median length of treatment 6 cycles - each cycle is 28 days (full range 2-12 cycles)
Population: Patients who received one full cycle of TMZ are evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
Number analyzed (Participants) | 17 | 15
Participants | 17 | 15

2. Primary Outcome: Duration of Response
Description: * Response and progression will be evaluated in this study using the updated response assessment criteria for high-grade gliomas: Response Assessment in Neuro-Oncology (RANO) working group guideline [JCO 28(11): 1963-1972, 2010].
  * The duration of overall response is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: Through completion of follow-up (estimated to be 30 months)
Population: Data was not collected for this outcome measure. Duration of response was never listed as an objective in the protocol; however it was erroneously mentioned in the statistical analysis section of the protocol and therefore was listed as a primary outcome measure in error as well.
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Patients Experiencing Grade 3 or 4 Lymphopenia, Thrombocytopenia, Neutropenia, Leukopenia, and Anemia in Each Group as Measured by Standard Blood Draws
Description: * Lymphopenia grade 3 is <500-200/mm^3 and grade 4 is <200/mm^3
  * Leukopenia grade 3 is <2000-1000/mm^3 and grade 4 is <1000/mm^3
  * Neutropenia grade 3 is <1000-500/mm^3 and grade 4 is <500/mm^3
  * Thrombocytopenia grade 3 is <50,000-25,000/mm^3 and grade 4 is <25,000/mm^3
  * Anemia grade 3 is <8.0-6.5 g/dL and grade 4 is <6.5 g/dL
Time Frame: Through completion of treatment (median length of treatment 6 cycles - each cycle is 28 days (full range 2-12 cycles)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
Number analyzed (Participants) | 22 | 20
Participants
  Lymphopenia | 2 | 0
  Thrombocytopenia | 1 | 0
  Neutropenia | 0 | 1
  Anemia | 1 | 0
  Leukopenia | 1 | 0

4. Secondary Outcome: Change in Quality of Life as Measured by FACT-Br Score - Physical Well-being Score
Description: 7-item questionnaire measuring over the past 7 days. Answers range from 0=not at all to 4=very much. Total score range is 0-28. A higher score indicates a lower physical well-being quality of life.
Time Frame: Baseline, beginning of each cycle (each cycle is 28 days), and 1 month after completion of treatment (up to 13 months, median length of treatment 6 cycles - each cycle is 28 days (full range 2-12 cycles))
Population: The number analyzed for each timepoint may be different from the overall number of participants analyzed if any participant did not complete the questionnaire at that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
Number analyzed (Participants) | 22 | 20
score on a scale
  Baseline | 6.23 (4.17) | 4.80 (4.27)
  Cycle 1: number analyzed (Participants) | 17 | 9
  Cycle 1 | 5.78 (4.96) | 4.00 (2.83)
  Cycle 2: number analyzed (Participants) | 16 | 14
  Cycle 2 | 7.66 (6.92) | 8.32 (5.65)
  Cycle 3: number analyzed (Participants) | 15 | 13
  Cycle 3 | 7.33 (5.67) | 7.69 (5.31)
  Cycle 4: number analyzed (Participants) | 14 | 12
  Cycle 4 | 6.18 (4.09) | 5.53 (4.74)
  Cycle 5: number analyzed (Participants) | 11 | 11
  Cycle 5 | 5.27 (4.54) | 7.03 (5.80)
  Cycle 6: number analyzed (Participants) | 11 | 7
  Cycle 6 | 4.64 (3.44) | 5.71 (5.59)
  Cycle 7: number analyzed (Participants) | 7 | 7
  Cycle 7 | 4.71 (4.19) | 3.00 (2.71)
  Cycle 8: number analyzed (Participants) | 6 | 6
  Cycle 8 | 3.83 (4.36) | 3.50 (4.14)
  Cycle 9: number analyzed (Participants) | 6 | 5
  Cycle 9 | 6.83 (4.62) | 4.00 (4.64)
  Cycle 10: number analyzed (Participants) | 6 | 4
  Cycle 10 | 5.35 (4.65) | 2.00 (1.63)
  Cycle 11: number analyzed (Participants) | 5 | 4
  Cycle 11 | 5.60 (5.59) | 2.00 (1.41)
  Cycle 12: number analyzed (Participants) | 4 | 3
  Cycle 12 | 4.50 (5.92) | 2.00 (1.00)
  End of treatment: number analyzed (Participants) | 16 | 13
  End of treatment | 5.19 (4.58) | 5.46 (3.82)

5. Secondary Outcome: Change in Quality of Life as Measured by FACT-Br Score - Social/Family Well-being Score
Description: 7-item questionnaire measuring over the past 7 days. Answers range from 0=not at all to 4=very much. Total score range 0-28. A higher score indicates a higher social/family well-being quality of life.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
Number analyzed (Participants) | 22 | 20
score on a scale
  Baseline | 24.10 (4.09) | 22.94 (3.98)
  Cycle 1: number analyzed (Participants) | 17 | 9
  Cycle 1 | 24.29 (4.13) | 22.59 (4.52)
  Cycle 2: number analyzed (Participants) | 16 | 14
  Cycle 2 | 22.45 (7.32) | 23.12 (4.18)
  Cycle 3: number analyzed (Participants) | 15 | 13
  Cycle 3 | 23.14 (5.93) | 22.26 (5.67)
  Cycle 4: number analyzed (Participants) | 14 | 12
  Cycle 4 | 23.21 (3.71) | 23.06 (4.78)
  Cycle 5: number analyzed (Participants) | 11 | 11
  Cycle 5 | 22.91 (4.72) | 22.30 (5.59)
  Cycle 6: number analyzed (Participants) | 11 | 7
  Cycle 6 | 22.44 (5.41) | 23.05 (5.13)
  Cycle 7: number analyzed (Participants) | 7 | 7
  Cycle 7 | 20.95 (6.31) | 24.86 (2.86)
  Cycle 8: number analyzed (Participants) | 6 | 6
  Cycle 8 | 22.78 (3.15) | 22.47 (4.26)
  Cycle 9: number analyzed (Participants) | 6 | 5
  Cycle 9 | 22.25 (4.40) | 22.52 (4.92)
  Cycle 10: number analyzed (Participants) | 6 | 4
  Cycle 10 | 22.94 (5.56) | 23.25 (2.63)
  Cycle 11: number analyzed (Participants) | 5 | 4
  Cycle 11 | 23.77 (3.09) | 26.08 (2.01)
  Cycle 12: number analyzed (Participants) | 4 | 3
  Cycle 12 | 24.00 (2.94) | 24.39 (1.99)
  End of treatment: number analyzed (Participants) | 17 | 15
  End of treatment | 21.95 (4.21) | 22.73 (4.38)

6. Secondary Outcome: Change in Quality of Life as Measured by FACT-Br Score - Emotional Well-being Score
Description: 6-item questionnaire measuring over the past 7 days. Answers range from 0=not at all to 4=very much. Total score range 0-24. A higher score indicates a lower emotional well-being quality of life.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
Number analyzed (Participants) | 22 | 20
score on a scale
  Baseline | 6.72 (3.72) | 7.60 (3.19)
  Cycle 1: number analyzed (Participants) | 17 | 9
  Cycle 1 | 6.69 (4.69) | 8.11 (2.85)
  Cycle 2: number analyzed (Participants) | 16 | 13
  Cycle 2 | 6.06 (4.82) | 6.77 (2.10)
  Cycle 3: number analyzed (Participants) | 15 | 13
  Cycle 3 | 6.63 (3.48) | 6.92 (2.14)
  Cycle 4: number analyzed (Participants) | 14 | 12
  Cycle 4 | 7.04 (3.25) | 5.47 (2.70)
  Cycle 5: number analyzed (Participants) | 11 | 11
  Cycle 5 | 6.68 (1.82) | 5.36 (2.01)
  Cycle 6: number analyzed (Participants) | 11 | 7
  Cycle 6 | 6.23 (3.45) | 5.57 (1.51)
  Cycle 7: number analyzed (Participants) | 7 | 7
  Cycle 7 | 7.29 (2.56) | 5.14 (2.73)
  Cycle 8: number analyzed (Participants) | 6 | 6
  Cycle 8 | 5.50 (3.15) | 5.67 (1.51)
  Cycle 9: number analyzed (Participants) | 6 | 5
  Cycle 9 | 7.33 (2.73) | 4.70 (1.99)
  Cycle 10: number analyzed (Participants) | 6 | 4
  Cycle 10 | 6.08 (3.58) | 5.25 (1.71)
  Cycle 11: number analyzed (Participants) | 5 | 4
  Cycle 11 | 8.60 (3.21) | 5.50 (1.91)
  Cycle 12: number analyzed (Participants) | 4 | 3
  Cycle 12 | 6.25 (2.22) | 8.33 (1.53)
  End of treatment: number analyzed (Participants) | 16 | 13
  End of treatment | 5.44 (3.22) | 5.62 (2.40)

7. Secondary Outcome: Change in Quality of Life as Measured by FACT-Br Score - Functional Well-being Score
Description: 7-item questionnaire measuring over the past 7 days. Answers range from 0=not at all to 4=very much. Total score range 0-28. A higher score indicates a higher emotional well-being quality of life.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
Number analyzed (Participants) | 22 | 20
score on a scale
  Baseline | 18.19 (6.39) | 16.35 (7.06)
  Cycle 1: number analyzed (Participants) | 17 | 9
  Cycle 1 | 18.71 (7.09) | 15.89 (7.59)
  Cycle 2: number analyzed (Participants) | 16 | 14
  Cycle 2 | 15.94 (8.68) | 16.11 (7.17)
  Cycle 3: number analyzed (Participants) | 15 | 13
  Cycle 3 | 16.37 (5.59) | 17.69 (5.86)
  Cycle 4: number analyzed (Participants) | 14 | 12
  Cycle 4 | 17.75 (6.82) | 18.78 (6.93)
  Cycle 5: number analyzed (Participants) | 11 | 11
  Cycle 5 | 17.32 (7.23) | 19.27 (7.86)
  Cycle 6: number analyzed (Participants) | 11 | 7
  Cycle 6 | 18.64 (7.66) | 20.00 (7.28)
  Cycle 7: number analyzed (Participants) | 7 | 7
  Cycle 7 | 18.71 (6.34) | 23.57 (5.77)
  Cycle 8: number analyzed (Participants) | 6 | 6
  Cycle 8 | 18.50 (7.18) | 21.00 (5.59)
  Cycle 9: number analyzed (Participants) | 6 | 5
  Cycle 9 | 17.00 (5.66) | 20.00 (6.89)
  Cycle 10: number analyzed (Participants) | 6 | 4
  Cycle 10 | 14.58 (8.48) | 25.00 (3.16)
  Cycle 11: number analyzed (Participants) | 5 | 4
  Cycle 11 | 18.80 (4.60) | 23.50 (4.12)
  Cycle 12: number analyzed (Participants) | 4 | 3
  Cycle 12 | 17.50 (6.24) | 23.33 (6.43)
  End of treatment: number analyzed (Participants) | 16 | 13
  End of treatment | 17.13 (8.24) | 18.54 (6.73)

8. Secondary Outcome: Median Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Time Frame: Through completion of follow-up (median length of follow-up 568.5 days, full range 1-1134 days)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
Number analyzed (Participants) | 22 | 20
months | 11.5978 [7.1952 to 29.6680] | 8.1809 [3.1869 to NA] — If fewer than half of the group have not experienced progression then upper 95% CI cannot be calculated.

9. Secondary Outcome: Median Overall Survival
Time Frame: Through completion of follow-up (median length of follow-up 568.5 days, full range 1-1134 days)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
Number analyzed (Participants) | 22 | 20
months | 26.9739 [10.6121 to 44.3869] | 17.1831 [8.3451 to NA] — If fewer than half of the group have not experienced death then upper 95% CI cannot be calculated.

10. Secondary Outcome: Comparison of Sleep Questionnaire in Participants Receiving Temozolomide in the Morning Versus Participants Receiving Temozolomide in the Evening
Description: Sleep Questionnaire - 1 yes/no question of "do you have problems getting to sleep or staying asleep?"
Time Frame: as for outcome 4
Population: Sleep questionnaires were only collected on 6 patients in each arm. If one of the 12 patients didn't complete a sleep questionnaire then they are not included in that timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
Number analyzed (Participants) | 6 | 6
Participants
  Baseline: Yes | 2 | 4
  Baseline: No | 4 | 2
  Cycle 1: number analyzed (Participants) | 4 | 5
  Cycle 1: Yes | 2 | 3
  Cycle 1: No | 2 | 2
  Cycle 2: number analyzed (Participants) | 4 | 5
  Cycle 2: Yes | 1 | 2
  Cycle 2: No | 3 | 3
  Cycle 3: number analyzed (Participants) | 4 | 5
  Cycle 3: Yes | 2 | 2
  Cycle 3: No | 2 | 3
  Cycle 4: number analyzed (Participants) | 4 | 5
  Cycle 4: Yes | 1 | 0
  Cycle 4: No | 3 | 5
  Cycle 5: number analyzed (Participants) | 2 | 5
  Cycle 5: Yes | 1 | 1
  Cycle 5: No | 1 | 4
  Cycle 6: number analyzed (Participants) | 3 | 3
  Cycle 6: Yes | 1 | 0
  Cycle 6: No | 2 | 3
  Cycle 7: number analyzed (Participants) | 3 | 1
  Cycle 7: Yes | 1 | 0
  Cycle 7: No | 2 | 1
  Cycle 8: number analyzed (Participants) | 2 | 1
  Cycle 8: Yes | 0 | 0
  Cycle 8: No | 2 | 1
  Cycle 9: number analyzed (Participants) | 2 | 1
  Cycle 9: Yes | 2 | 0
  Cycle 9: No | 0 | 1
  Cycle 10: number analyzed (Participants) | 2 | 1
  Cycle 10: Yes | 2 | 0
  Cycle 10: No | 0 | 1
  Cycle 11: number analyzed (Participants) | 2 | 1
  Cycle 11: Yes | 1 | 0
  Cycle 11: No | 1 | 1
  Cycle 12: number analyzed (Participants) | 2 | 1
  Cycle 12: Yes | 1 | 0
  Cycle 12: No | 1 | 1
  End of Treatment: number analyzed (Participants) | 3 | 6
  End of Treatment: Yes | 1 | 0
  End of Treatment: No | 2 | 6

11. Secondary Outcome: Comparison of Sleep Questionnaire in Participants Receiving Temozolomide in the Morning Versus Participants Receiving Temozolomide in the Evening
Description: - Sleep Questionnaire:
  * Difficulty falling asleep/difficulty staying asleep/problem waking up too early: Answers range from 0=none, mild=1, moderate=2, severe=3, very=4.
  * How satisfied or dissatisfied are you with your current sleeping pattern question: Answers range from 0=very satisfied to 4=very dissatisfied.
  * To what extent do you consider your sleep problem to interfere with your daily functioning question: Answers range from 0=not at all interfering, 1=a little, 2=somewhat, 3=much, 4=very much interfering.
  * How noticeable to others do you think your sleep problem is in terms of impairing the quality of your life question: Answers range from 0=not at all noticeable, 1=barely, 2 = somewhat, 3 =much, 4=very noticeable.
  * How worried or distressed are you about your current sleep problem question: Answers range from 0=not at all=0, 1=a little, 2=somewhat, 3=much, 4=very much.
Time Frame: as for outcome 4
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Temozolomide Morning BASELINE; Arm 1: Temozolomide Morning CYCLE 1; Arm 1: Temozolomide Morning CYCLE 2; Arm 1: Temozolomide Morning CYCLE 3; Arm 1: Temozolomide Morning CYCLE 4; Arm 1: Temozolomide Morning CYCLE 5; Arm 1: Temozolomide Morning CYCLE 6; Arm 1: Temozolomide Morning CYCLE 7; Arm 1: Temozolomide Morning CYCLE 8; Arm 1: Temozolomide Morning CYCLE 9; Arm 1: Temozolomide Morning CYCLE 10; Arm 1: Temozolomide Morning CYCLE 11; Arm 1: Temozolomide Morning CYCLE 12; Arm 1: Temozolomide Morning END OF TREATMENT: -Temozolomide will be given as per standard of care. Typical dosing is 150 to 200 mg/m^2 on Days 1 through 5 of a 28-day treatment cycle. Patients will be randomized to take their temozolomide doses in the morning (before 10:00).
- Arm 2: Temozolomide Evening BASELINE; Arm 2: Temozolomide Evening CYCLE 1; Arm 2: Temozolomide Evening CYCLE 2; Arm 2: Temozolomide Evening CYCLE 3; Arm 2: Temozolomide Evening CYCLE 4; Arm 2: Temozolomide Evening CYCLE 5; Arm 2: Temozolomide Evening CYCLE 6; Arm 2: Temozolomide Evening CYCLE 7; Arm 2: Temozolomide Evening CYCLE 8; Arm 2: Temozolomide Evening CYCLE 9; Arm 2: Temozolomide Evening CYCLE 10; Arm 2: Temozolomide Evening CYCLE 11; Arm 2: Temozolomide Evening CYCLE 12; Arm 2: Temozolomide Evening END OF TREATMENT: -Temozolomide will be given as per standard of care. Typical dosing is 150 to 200 mg/m2 on Days 1 through 5 of a 28-day treatment cycle. Patients will be randomized to take their temozolomide doses in the evening (after 20:00).
Arm/Group | Arm 1: Temozolomide Morning BASELINE | Arm 2: Temozolomide Evening BASELINE | Arm 1: Temozolomide Morning CYCLE 1 | Arm 2: Temozolomide Evening CYCLE 1 | Arm 1: Temozolomide Morning CYCLE 2 | Arm 2: Temozolomide Evening CYCLE 2 | Arm 1: Temozolomide Morning CYCLE 3 | Arm 2: Temozolomide Evening CYCLE 3 | Arm 1: Temozolomide Morning CYCLE 4 | Arm 2: Temozolomide Evening CYCLE 4 | Arm 1: Temozolomide Morning CYCLE 5 | Arm 2: Temozolomide Evening CYCLE 5 | Arm 1: Temozolomide Morning CYCLE 6 | Arm 2: Temozolomide Evening CYCLE 6 | Arm 1: Temozolomide Morning CYCLE 7 | Arm 2: Temozolomide Evening CYCLE 7 | Arm 1: Temozolomide Morning CYCLE 8 | Arm 2: Temozolomide Evening CYCLE 8 | Arm 1: Temozolomide Morning CYCLE 9 | Arm 2: Temozolomide Evening CYCLE 9 | Arm 1: Temozolomide Morning CYCLE 10 | Arm 2: Temozolomide Evening CYCLE 10 | Arm 1: Temozolomide Morning CYCLE 11 | Arm 2: Temozolomide Evening CYCLE 11 | Arm 1: Temozolomide Morning CYCLE 12 | Arm 2: Temozolomide Evening CYCLE 12 | Arm 1: Temozolomide Morning END OF TREATMENT | Arm 2: Temozolomide Evening END OF TREATMENT
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 5 | 5 | 5 | 5 | 4 | 5 | 4 | 5 | 3 | 4 | 3 | 1 | 2 | 1 | 3 | 1 | 3 | 1 | 2 | 1 | 2 | 1 | 3 | 6
Participants
  Difficulty falling asleep: number analyzed (Participants) | 6 | 6 | 4 | 5 | 5 | 5 | 5 | 5 | 4 | 5 | 4 | 5 | 3 | 4 | 3 | 1 | 2 | 1 | 3 | 1 | 3 | 1 | 2 | 1 | 2 | 1 | 3 | 6
  Difficulty falling asleep: 0 | 3 | 1 | 2 | 1 | 3 | 2 | 3 | 0 | 2 | 4 | 2 | 4 | 1 | 3 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 2
  Difficulty falling asleep: 1 | 1 | 2 | 1 | 1 | 2 | 1 | 0 | 4 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 3
  Difficulty falling asleep: 2 | 2 | 1 | 1 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  Difficulty falling asleep: 3 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Difficulty falling asleep: 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Difficulty staying asleep: number analyzed (Participants) | 6 | 6 | 4 | 5 | 5 | 5 | 5 | 5 | 4 | 5 | 4 | 5 | 3 | 4 | 3 | 1 | 2 | 1 | 3 | 1 | 3 | 1 | 2 | 1 | 2 | 1 | 3 | 6
  Difficulty staying asleep: 0 | 4 | 2 | 2 | 2 | 3 | 0 | 3 | 0 | 3 | 3 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 2
  Difficulty staying asleep: 1 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 4 | 0 | 1 | 2 | 3 | 1 | 3 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 3
  Difficulty staying asleep: 2 | 2 | 1 | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Difficulty staying asleep: 3 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Difficulty staying asleep: 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Problem waking up too early: number analyzed (Participants) | 6 | 6 | 4 | 5 | 5 | 5 | 5 | 5 | 4 | 5 | 4 | 5 | 3 | 4 | 3 | 1 | 2 | 1 | 3 | 1 | 3 | 1 | 2 | 1 | 2 | 1 | 3 | 6
  Problem waking up too early: 0 | 3 | 1 | 3 | 1 | 3 | 1 | 4 | 1 | 2 | 1 | 1 | 4 | 2 | 3 | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 2 | 1 | 2 | 3
  Problem waking up too early: 1 | 1 | 2 | 0 | 1 | 2 | 3 | 0 | 1 | 1 | 3 | 3 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  Problem waking up too early: 2 | 2 | 3 | 1 | 3 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Problem waking up too early: 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Problem waking up too early: 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  How satisfied or dissatisfied are you with your current sleeping pattern?: number analyzed (Participants) | 6 | 6 | 4 | 5 | 5 | 5 | 5 | 5 | 4 | 5 | 4 | 5 | 3 | 4 | 3 | 1 | 2 | 1 | 3 | 1 | 3 | 1 | 2 | 1 | 2 | 1 | 3 | 6
  How satisfied or dissatisfied are you with your current sleeping pattern?: 0 | 3 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 2
  How satisfied or dissatisfied are you with your current sleeping pattern?: 1 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 2 | 2 | 2 | 2 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0
  How satisfied or dissatisfied are you with your current sleeping pattern?: 2 | 3 | 3 | 2 | 3 | 1 | 1 | 1 | 2 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  How satisfied or dissatisfied are you with your current sleeping pattern?: 3 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  How satisfied or dissatisfied are you with your current sleeping pattern?: 4 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  To what extent do you consider your sleep problem to interfere with your daily functioning?: number analyzed (Participants) | 6 | 6 | 4 | 5 | 5 | 5 | 5 | 5 | 4 | 5 | 4 | 5 | 3 | 4 | 3 | 1 | 2 | 1 | 3 | 1 | 3 | 1 | 2 | 1 | 2 | 1 | 3 | 6
  To what extent do you consider your sleep problem to interfere with your daily functioning?: 0 | 3 | 2 | 1 | 2 | 3 | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 0
  To what extent do you consider your sleep problem to interfere with your daily functioning?: 1 | 1 | 2 | 0 | 2 | 0 | 4 | 1 | 2 | 1 | 3 | 1 | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 4
  To what extent do you consider your sleep problem to interfere with your daily functioning?: 2 | 2 | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  To what extent do you consider your sleep problem to interfere with your daily functioning?: 3 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  To what extent do you consider your sleep problem to interfere with your daily functioning?: 4 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  How noticeable to others is your sleep problem is in terms of impairing the quality of your life: number analyzed (Participants) | 6 | 6 | 4 | 5 | 5 | 5 | 5 | 5 | 4 | 5 | 4 | 5 | 3 | 4 | 3 | 1 | 2 | 1 | 3 | 1 | 3 | 1 | 2 | 1 | 2 | 1 | 3 | 6
  How noticeable to others is your sleep problem is in terms of impairing the quality of your life: 0 | 3 | 0 | 1 | 0 | 2 | 2 | 2 | 0 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 2
  How noticeable to others is your sleep problem is in terms of impairing the quality of your life: 1 | 1 | 2 | 0 | 2 | 0 | 2 | 1 | 3 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 2
  How noticeable to others is your sleep problem is in terms of impairing the quality of your life: 2 | 2 | 2 | 3 | 1 | 3 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  How noticeable to others is your sleep problem is in terms of impairing the quality of your life: 3 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  How noticeable to others is your sleep problem is in terms of impairing the quality of your life: 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  How worried or distressed are you about your current sleep problem?: number analyzed (Participants) | 6 | 6 | 4 | 5 | 5 | 5 | 5 | 5 | 4 | 5 | 4 | 5 | 3 | 4 | 3 | 1 | 2 | 1 | 3 | 1 | 3 | 1 | 2 | 1 | 2 | 1 | 3 | 6
  How worried or distressed are you about your current sleep problem?: 0 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 3 | 3 | 2 | 3 | 1 | 4 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 5
  How worried or distressed are you about your current sleep problem?: 1 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 1
  How worried or distressed are you about your current sleep problem?: 2 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  How worried or distressed are you about your current sleep problem?: 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  How worried or distressed are you about your current sleep problem?: 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Mean Circadian Amplitude
Description: * The ActTrust Condor Instrument watches are wrist actimetry/accelerometers. Patients will wear an accelerometer on their wrist to measure activity level during the day and at night until two months after the end of treatment.
  * Circadian amplitude, refers to the difference between the highest and lowest points of a circadian rhythm over a 24-hour cycle, is typically measured in the units of the rhythm being quantified.
  * The circadian mean amplitude was calculated per day for each patient with the mean and standard deviation reported across all days for each individual patient.
Time Frame: From start of treatment through 2 months after end of treatment (median length 100 days, full range 78-240 days)
Population: Actimetry data was only collected on 6 participants.
Measure: Mean (Standard Deviation); unit: counts/minute
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
Number analyzed (Participants) | 2 | 4
counts/minute
  AM Patient #1: number analyzed (Participants) | 1 | 0
  AM Patient #1 | 0.78 (0.02) |
  AM Patient #2: number analyzed (Participants) | 1 | 0
  AM Patient #2 | 0.78 (0.01) |
  PM Patient #1: number analyzed (Participants) | 0 | 1
  PM Patient #1 |  | 0.81 (0.01)
  PM Patient #2: number analyzed (Participants) | 0 | 1
  PM Patient #2 |  | 0.78 (0.01)
  PM Patient #3: number analyzed (Participants) | 0 | 1
  PM Patient #3 |  | 0.77 (0.02)
  PM Patient #4: number analyzed (Participants) | 0 | 1
  PM Patient #4 |  | 0.81 (0.01)

13. Secondary Outcome: Mean Sleep Regularity Index (SRI)
Description: * The ActTrust Condor Instrument watches are wrist actimetry/accelerometers. Patients will wear an accelerometer on their wrist to measure activity level during the day and at night until two months after the end of treatment.
  * Sleep regularity index (SRI) is the probability of being at rest, calculated per day for each patient. An SRI closer to 0 indicates irregular sleep patterns (i.e., more variable day to day), while values closer to 1 indicate regular sleep patterns. The SRI index scale is 0~1.
  * The SRI was calculated per day for each patient with the mean and standard deviation reported across all days for each individual patient.
Time Frame: From start of treatment through 2 months after end of treatment (median length 100 days, full range 78-240 days)
Population: Actimetry data was only collected on 6 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
Number analyzed (Participants) | 2 | 4
units on a scale
  AM Patient #1: number analyzed (Participants) | 1 | 0
  AM Patient #1 | 0.70 (0.09) |
  AM Patient #2: number analyzed (Participants) | 1 | 0
  AM Patient #2 | 0.79 (0.8) |
  PM Patient #1: number analyzed (Participants) | 0 | 1
  PM Patient #1 |  | 0.82 (0.09)
  PM Patient #2: number analyzed (Participants) | 0 | 1
  PM Patient #2 |  | 0.69 (0.10)
  PM Patient #3: number analyzed (Participants) | 0 | 1
  PM Patient #3 |  | 0.68 (0.08)
  PM Patient #4: number analyzed (Participants) | 0 | 1
  PM Patient #4 |  | 0.82 (0.11)

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from start of treatment through completion of follow-up (median length of follow-up 568.5 days, full range 1-1134 days) Adverse events were collected from start of treatment through end of treatment visit (median length of treatment 6 cycles - each cycle is 28 days (full range 2-12 cycles).
Description: Only grade 3 or higher hematologic adverse events were collected along with all serious adverse events.
Arm/Group | Arm 1: Temozolomide Morning | Arm 2: Temozolomide Evening
All-Cause Mortality (participants affected / at risk) | 7/22 | 6/20
Serious Adverse Events (participants affected / at risk) | 6/22 | 5/20
Other Adverse Events (participants affected / at risk) | 4/22 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Temozolomide Morning (N=22) | Arm 2: Temozolomide Evening (N=20)
Aspartate aminotransferase increased (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Death due to disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Temozolomide Morning (N=22) | Arm 2: Temozolomide Evening (N=20)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT02781792/Prot_SAP_000.pdf